CLINICAL TRIAL: NCT05503004
Title: The Second Affilliated Hospital of Zhejiang University, School of Medicine
Brief Title: Prehabilitation in Adult Patients Following Selective Cardiac Surgery: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20220630
Record Dates: First submitted 2022-08-01; First posted 2022-08-16 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-06

CONDITIONS: Enhanced Recovery; Prehabilitation; Cardiac Surgery
MeSH Terms: interventions — Preoperative Exercise; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): comprehensive prehabilitation program including supervised exercise., mindfulness and nutrition assessment.
  Interventions: Behavioral: Prehabilitation
- Standard care (Active Comparator): Standard care before surgery
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Prehabilitation — 10 min exercise, 5 min respiratory mindfulness, and preoperative nutrition assessment.
  Arms: Intervention group
Behavioral: Standard care — Standard care before surgery
  Arms: Standard care

SUMMARY:
Aim: To determine the impact of an evidence-based comprehensive prehabilitation (EBCPrehab) program on pre- and postoperative capacity, functional capacity and health related quality of life (HRQoL) in patients awaiting elective coronary artery bypass graft surgery (CABG) or valvular surgery. Design: A single-center randomized controlled trail. SUBJECTS: Overall 160 preoperative elective cardiac surgery patients will be randomly assigned to an intervention or control group. Intervention: one-week EBCPrehab intervention, including supervised exercise, mindfulness and nutrition assessment. Control group: usual care. Main measures: At baseline, one day before surgery, three days after surgery and before discharge. The following measurements will be performed: six-minute walk test, ICU delirium, health related quality of life and flow state.

DETAILED DESCRIPTION:
Enhanced recovery improves the quality of recovery following cardiac surgery, while the evidence of prehabilitation is still limited. We hypothesize that the implementation of a comprehensive prehabilitation program, including physical, mental and nutrition support could optimize the postoperative outcomes during hospital stay.

A randomized controlled study of patients undergoing cardiac surgery with prehabilitation approach, is designed to compare patient outcomes. The samples will be collected from hospital registration and the invention will be conducted before surgery. During the 5-day prehabilitation intervention, patients will receive exercises, mindfulness and nutrition risk assessment. After surgery, the 6-minute walk test, delirium assessment, flow state and health related quality of life will be assessed to explore the effects of prehabilitation on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients awaiting selective coronary artery bypass graft surgery (CABG) or valvular surgery

Exclusion Criteria:

* Disability, severe psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative physical function | up to 1 week
  6-minute walk test distance in meters
Postoperative physical function | up to 2 weeks
  6-minute walk test distance in meters

SECONDARY OUTCOMES:
ICU delirium | Up to 5 days
  Assessed by nurses every shift using the Confusion Assessment Method of the Intensive Care Unit -7 (CAM-ICU-7). The CAM-ICU-7 score ranges from 0-7 with 7 being most severe.
Health related quality of life | up to 4 weeks
  Using the The EuroQol 5 Dimension 5 Level (EQ-5D-5L). The EQ-5D-5L defines health conditions based on five dimensions (e.g. mobility, self-care, usual activities, pain/discomfort, and anxiety/depression).
Flow State | up to 2 weeks
  Using the The Flow State Scale for Occupational Tasks (FSSOT). The total score ranges from 14 to 98 points. The high score is considered to indicate the strong flow state in performing a specific task.
Postoperative delirium | Up to 2 weeks
  Assessed by nurses every shift using the 4AT Rapid clinical test for delirium. The 4AT is scored from 0-12. A score of 4 or more suggests delirium.
Gut microbiome diversity | up to 2 weeks
  Stool collection and 16s RNA analysis
Short chain fatty acids (SCFAs) | up to 2 weeks
  Stool collection and SCFAs quantitative analysis

CONTACTS AND LOCATIONS:
Overall Officials: Wen Gao, PhD, Principal Investigator — Zhejiang University
Locations (1):
- Second Affiliated hospital of Zhejiang university School of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao W, Li H, Chen Y, Zhang Y, Zhang M, Jin J. Effectiveness of a short-term multimodal prehabilitation program in adult patients awaiting selective cardiac surgery: study protocol for an open-label, pilot, randomized controlled trial. Front Cardiovasc Med. 2023 Jun 30;10:1201737. doi: 10.3389/fcvm.2023.1201737. eCollection 2023. PMID 37456818